CLINICAL TRIAL: NCT02806102
Title: Cardiovascular Risk and Identification of Potential High-risk Population in Korean Patients With Acute Myocardial Infarction II (COREA-AMI II)
Brief Title: CardiOvascular Risk and idEntificAtion of Potential High-risk Population in Acute Myocardial Infarction II (COREA-AMI II)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: The Catholic University of Korea (Other); Chonnam National University (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Kiyuk Chang, Chief of the Division of Cardiology, Seoul St. Mary's Hospital
Other Study IDs: XC15RSMI0089K
Record Dates: First submitted 2016-05-31; First posted 2016-06-20 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: Acute Myocardial Infarction; Percutaneous Coronary Intervention; Major Adverse Cardiovascular Events; Bleeding
MeSH Terms: conditions — Hemorrhage | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years

GROUPS / COHORTS (2):
- High-risk: Acute myocardial infarction treated with percutaneous coronary intervention and/or long-term use of dual-antiplatelet therapy and have at least one of the following risk factors:
  * Age ≥ 65 years
  * Diabetes mellitus requiring medication
  * Documented history of a second prior presumed spontaneous MI (>1 year ago)
  * Documented history of angiographic evidence of multivessel coronary artery disease
  * Chronic, non-end stage renal dysfunction
  Interventions: Procedure: Percutaneous coronary intervention; Drug: Dual-antiplatelet therapy
- Low-risk: Acute myocardial infarction treated with percutaneous coronary intervention and/or long-term use of dual-antiplatelet therapy and have none of the pre-specified risk factors
  Interventions: Procedure: Percutaneous coronary intervention; Drug: Dual-antiplatelet therapy

INTERVENTIONS:
Procedure: Percutaneous coronary intervention — Percutaneous coronary intervention
  Other Names: PCI
  Groups: High-risk
Drug: Dual-antiplatelet therapy — Dual AntiPlatelet Therapy
  Other Names: DAPT
  Groups: High-risk
Procedure: Percutaneous coronary intervention — Percutaneous coronary intervention
  Other Names: PCI
  Groups: Low-risk
Drug: Dual-antiplatelet therapy — Dual AntiPlatelet Therapy
  Other Names: DAPT
  Groups: Low-risk

SUMMARY:
This study is intended to provide contemporary data on the residual cardiovascular risk in all consecutive patients with acute myocardial infarction, especially in patients who survived stably within one-year after percutaneous coronary intervention.

In addition, this study will identify which baseline clinical, angiographic, or treatment factors are associated with residual cardiovascular risk and bleeding events

DETAILED DESCRIPTION:
COREA-AMI registry was conducted previously (NCT02385682) and enrolled consecutive all patient with acute myocardial infarction who were treated with percutaneous coronary intervention from Jan 2004 to Dec 2009.

COREA-AMI II registry extend the enrollment period to Aug 2014 and the follow-up period to Jun 2016.

All consecutive acute myocardial infarction patients had been enrolled prospectively in prior registries of each university hospitals. Eight hospitals of the Catholic University of Korea already have web-based coronary intervention registry (NCT01239914). And Cheonnam University Hospital is one of leading hospitals to design and manage the web-based previous Korean nationwide myocardial infarction registry, the Korea Acute Myocardial Infarction Registry (KAMIR) (http://www.kamir.or.kr/).

Using these previous data, the current registry update new clinical and angiographic variables and assess long-term clinical follow-up data retrospectively. All data were collected on web-based system after eliminating personal information. (http://www.ecrf.kr/coreaami/)

All data are going to be sealed with code by Clinical Research Coordinating Center of the Catholic University of Korea and to be managed and analyzed by independent statistics perssonels.

Cardiovascular center with high-volume percutaneous coronary intervention of following hospitals were participated.

* Seoul St. Mary's Hospital, Seoul, South Korea
* Yeoido St. Mary's Hospital, Seoul, South Korea
* Uijongbu St. Mary's Hospital, Gyeonggi-do, South Korea
* St. Paul Hospital, Seoul, South Korea
* Bucheon St. Mary's Hospital, Gyeonggi-do, South Korea
* Incheon St. Mary's Hospital, Incheon, South Korea
* St. Vincent Hospital, Gyeonggi-do, South Korea
* Deajon St. Mary's Hospital, Daejeon, South Korea
* Cheonnam University Hospital, Gwangju, South Korea

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction who were treated with percutaneous coronary intervention using stents

Exclusion Criteria:

* Acute myocardial infarction who were treated with only balloon angioplasty
* Acute myocardial infarction who were managed by conservative strategy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute myocardial infarction who were treated with percutaneous coronary intervention
Sampling Method: Non-Probability Sample
Enrollment: 13000 (Estimated)
Dates: Start 2004-01; Primary Completion 2017-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of cardiovascular events | 5 years
  Cardiac death, nonfatal myocardial infarction, or nonfatal stroke

SECONDARY OUTCOMES:
Cumulative incidence of all-cause death | 5 years
Cumulative incidence of cardiac death | 5 years
Cumulative incidence of nonfatal myocardial infarction | 5 years
Cumulative incidence of nonfatal stroke | 5 years
Cumulative incidence of target lesion revascularization | 5 years
Cumulative incidence of target vessel revascularization | 5 years
Cumulative incidence of non-target vessel revascularization | 5 years
Cumulative incidence of definite/Probable stent thrombosis | 5 years
Cumulative incidence of hospitalization for heart failure | 5 years
Cumulative incidence of bleeding defined as the Bleeding Academic Research Consortium definitions type 2, 3, and 5 | 5 years
Bleeding defined as the thrombolysis In Myocardial Infarction major/minor | 5 years
Cumulative incidence of major adverse cardiac and cerebrovascular events | 5 years
  All-cause death, nonfatal myocardial infarction, nonfatal stroke, or any revascularization

OTHER OUTCOMES:
Cumulative incidence of cardiovascular events beyond first year after percutaneous coronary intervention | From 1 year up to 5 years after percutaneous coronary intervention
  Cardiac death, nonfatal myocardial infarction, or nonfatal stroke

CONTACTS AND LOCATIONS:
Overall Officials: Kiyuk Chang, MD, PhD, Principal Investigator — Seoul St. Mary's Hospital; Youngkeun Ahn, MD, PhD, Study Director — Chonnam National University Hospital
Locations (2):
- South Korea (2):
  - Chonnam National University Hospital, Gwangju
  - Seoul St. Mary's Hospital, The Catholic University of Korea, Seoul

REFERENCES:
- [Derived] Kim SH, Lee W, Choo EH, Lee KY, Hwang BH, Choi IJ, Lee JM, Yoo KD, Park MW, Park CS, Kim HY, Kim MC, Ahn Y, Chang K. Long-term outcomes of premature acute myocardial infarction: impact of multivessel disease. Coron Artery Dis. 2026 Jan 20. doi: 10.1097/MCA.0000000000001613. Online ahead of print. PMID 41555573
- [Derived] Kim SH, Choo EH, Kang J, Lee JM, Yoo KD, Park MW, Park CS, Kim HY, Kim MC, Ahn Y, Chang K, Kim HS. The efficacy and safety of prasugrel in acute coronary syndrome: a propensity-matched Korean cohort study focused on age and weight of patients. BMC Cardiovasc Disord. 2025 Nov 26;25(1):888. doi: 10.1186/s12872-025-05263-w. PMID 41299333
- [Derived] Kim S, Lee KY, Kim KA, Byeon J, Shin S, Hwang BH, Kim JJ, Choo EH, Kim CJ, Kyoung Sa Y, Park MW, Hyun S, Yoon AH, Ahn Y, Chang K. The role of serum uric acid in survival prediction in patients with acute myocardial infarction accompanied by heart failure with preserved ejection fraction. Front Cardiovasc Med. 2025 Nov 10;12:1622275. doi: 10.3389/fcvm.2025.1622275. eCollection 2025. PMID 41293617
- [Derived] Kim KA, Kim SH, Lee KY, Yoon AH, Hwang BH, Choo EH, Kim JJ, Choi IJ, Kim CJ, Lim S, Park MW, Yoo KD, Jeon DS, Ahn Y, Jeong MH, Chang K. Predictors and Long-Term Clinical Impact of Heart Failure With Improved Ejection Fraction After Acute Myocardial Infarction. J Am Heart Assoc. 2024 Aug 20;13(16):e034920. doi: 10.1161/JAHA.124.034920. Epub 2024 Aug 19. PMID 39158557
- [Derived] Lee M, Lee K, Kim DW, Cho JS, Kim TS, Kwon J, Kim CJ, Park CS, Kim HY, Yoo KD, Jeon DS, Chang K, Kim MC, Jeong MH, Ahn Y, Park MW. Comparative Effectiveness of Long-Term Maintenance Beta-Blocker Therapy After Acute Myocardial Infarction in Stable, Optimally Treated Patients Undergoing Percutaneous Coronary Intervention. J Am Heart Assoc. 2023 Aug;12(15):e028976. doi: 10.1161/JAHA.122.028976. Epub 2023 Jul 26. PMID 37493020
- [Derived] Kim HY, Mok J, Kim JY, Jeon D, Her SH, Park MW, Kim DB, Park CS, Lee JM, Chang K, Jung WS, Ahn Y. Effect of Angiotensin Receptor Blocker Dose in Myocardial Infarction With Preserved Left Ventricular Systolic Function. J Cardiovasc Pharmacol. 2023 Jul 1;82(1):52-60. doi: 10.1097/FJC.0000000000001427. PMID 37019077
- [Derived] Ahn Y, Lee D, Choo EH, Choi IJ, Lim S, Lee KY, Hwang BH, Park MW, Lee JM, Park CS, Kim HY, Yoo KD, Jeon DS, Chung WS, Kim MC, Jeong MH, Ahn Y, Chang K. Association Between Bleeding and New Cancer Detection and the Prognosis in Patients With Myocardial Infarction. J Am Heart Assoc. 2022 Nov 15;11(22):e026588. doi: 10.1161/JAHA.122.026588. Epub 2022 Nov 8. PMID 36346059
- [Derived] Cho KH, Kim MC, Choo EH, Choi IJ, Lee SN, Park MW, Park CS, Kim HY, Kim CJ, Sim DS, Kim JH, Hong YJ, Jeong MH, Chang K, Ahn Y. Impact of Low Baseline Low-Density Lipoprotein Cholesterol on Long-Term Postdischarge Cardiovascular Outcomes in Patients With Acute Myocardial Infarction. J Am Heart Assoc. 2022 Sep 6;11(17):e025958. doi: 10.1161/JAHA.122.025958. Epub 2022 Aug 24. PMID 36000434
- [Derived] Lee M, Lee K, Kim DW, Cho JS, Kim TS, Kwon J, Kim CJ, Park CS, Kim HY, Yoo KD, Jeon DS, Chang K, Kim MC, Jeong MH, Ahn Y, Park MW. Relationship of Serial High-Sensitivity C-Reactive Protein Changes to Long-term Clinical Outcomes in Stabilised Patients After Myocardial Infarction. Can J Cardiol. 2022 Jan;38(1):92-101. doi: 10.1016/j.cjca.2021.10.007. Epub 2021 Nov 2. PMID 34737035